CLINICAL TRIAL: NCT00287066
Title: Open-Label Randomized Two-Way Crossover Pilot Study To Estimate The Effects Of Inhaled Versus IV Infusion Of Human Insulin With Regards To Glucose Disposal In Subjects With Type 1 Diabetes Mellitus
Brief Title: A Clinical Trial Assessing the Impact of Inhaled Insulin on Glucose Disposition
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A2171060
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

INTERVENTIONS:
Drug: Inhaled Human Insulin
Drug: Regular Human Insulin

SUMMARY:
To assess the impact of inhalation of insulin on glucose disposition in patients with type 1 diabetes

DETAILED DESCRIPTION:
The study was terminated on Oct. 28, 2007. The protocol was undergoing implementation and methodological issues with major revisions that qualified this trial as a new trial. Pfizer decided to cancel new trials because of the decision to withdraw Exubera due to lack of market performance and not for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 1

Exclusion Criteria:

* Asthma, COPD
* Smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
18F-labeled glucose uptake in muscle

SECONDARY OUTCOMES:
Glucose turnover overnight Insulin pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171060&StudyName=A+Clinical+Trial+Assessing+the+Impact+of+Inhaled+Insulin+on+Glucose+Disposition